CLINICAL TRIAL: NCT04533204
Title: Comparing Mnemonic Strategy With Spaced Retrieval Training in Patients With Mild Cognitive Impairment (B6366-W)
Brief Title: Mnemonic Strategy Versus Spaced Retrieval Training in Those With Mild Cognitive Impairment
Acronym: MST training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6366-W-1
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-11

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; cognitive training; memory training; dementia; Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Randomization to Mnemonic strategy or spaced retrieval training
Who Masked: Participant
Masking Description: Participants were informed they would receive one of two cognition oriented treatments but were unaware of the nature of the other intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mnemonic strategy training (Experimental): Training using mnemonic strategies
  Interventions: Behavioral: mnemonic strategy training
- Spaced retrieval training (Active Comparator): Training using spaced retrieval
  Interventions: Behavioral: spaced retrieval training

INTERVENTIONS:
Behavioral: mnemonic strategy training — training using mnemonic strategies
  Arms: Mnemonic strategy training
Behavioral: spaced retrieval training — training using spaced retrieval
  Arms: Spaced retrieval training

SUMMARY:
This study compared two active cognitive interventions to evaluate whether one improved memory more than the other in patients with mild cognitive impairment. Participants were randomized to either memory strategy training or spaced retrieval training and completed memory tests before and after 3 training sessions. Participants returned 1 month after treatment to see how well they remembered the learned information. Brain scans (functional MRI) were collected before and after the interventions to see if training changed the way brain regions were functioning.

DETAILED DESCRIPTION:
Individuals with MCI were randomized to 3 sessions of mnemonic strategy or spaced retrieval training that focused on object location associations. Across these training sessions, each group received 9 training trials for each of the 45 trained stimuli. Task-fMRI was acquired before and after training. Memory was again evaluated 1 month after the last training session. The primary outcome measure was memory for the "trained" stimuli while secondary outcome was accuracy for novel stimuli acquired outside of the MRI environment.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of MCI according to Petersen (2004) criteria, right handed

Exclusion Criteria:

* Diagnosis of other neurological condition,
* active drug/alcohol abuse/dependence,
* moderate-severe depression or other Axis I diagnoses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M. Hampstead, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mnemonic Strategy Training | Spaced Retrieval Training
Started | 29 | 30
Completed | 28 | 29
Not Completed | 1 | 1
Not completed — Unable to understand training instructions | 1 | 1

BASELINE CHARACTERISTICS:
Population: All diagnosed with amnestic MCI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mnemonic Strategy Training | Spaced Retrieval Training | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 participant in each group was removed due to inability to understand training instructions
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 7 | 12
    >=65 years | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 1 participant in each group removed due to inability to understand training instructions
  Years | 72.7 (8.3) | 70.5 (8.3) | 71.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant in each group removed due to inability to understand training instructions
  Participants
    Female | 10 | 14 | 24
    Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant in each group removed due to inability to understand training instructions
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 11 | 19
    White | 19 | 17 | 36
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percent of Correct Object Location Associations Assessed up to 1 Month Post-treatment
Description: Change in memory for 45 trained object location associations
Time Frame: up to 1 month after last training session
Measure: Mean (95% Confidence Interval); unit: percent correct
Arm/Group | Mnemonic Strategy Training | Spaced Retrieval Training
Number analyzed (Participants) | 28 | 29
percent correct | 80.0 [74.86 to 85.14] | 62.45 [57.4 to 67.51]
Statistical Analysis 1: Comparison: Mnemonic Strategy Training vs Spaced Retrieval Training; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = 18.47, 95% CI 2-sided [12.28 to 24.67]

2. Secondary Outcome: Change in Accuracy (vs. Baseline) on Novel Object Location Associations
Description: Change in accuracy for novel object location associations using a touchscreen task; distance measured in cm from actual location
Time Frame: up to 1 month after last training session
Population: Computer errors resulted in loss of data from the first 15 participants (7 MST, 8 SRT)
Measure: Mean (95% Confidence Interval); unit: error in centimeters
Arm/Group | Mnemonic Strategy Training | Spaced Retrieval Training
Number analyzed (Participants) | 21 | 21
error in centimeters | 6.1 [4.8 to 7.4] | 7.14 [5.84 to 8.44]
Statistical Analysis 1: Comparison: Mnemonic Strategy Training vs Spaced Retrieval Training; Test type: Superiority; p = .004, Mixed Models Analysis — Performance on cued recall (error scores); Mean Difference (Final Values) = 2.33, 95% CI 2-sided [.75 to 3.91]

ADVERSE EVENTS:
Arm/Group | Mnemonic Strategy Training | Spaced Retrieval Training
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No